CLINICAL TRIAL: NCT00047814
Title: A Multiple Rising-Dose Study of FK788 in Subjects With Chronic Hepatitis C Virus Infection
Brief Title: Study of FK788 in Subjects With Chronic Hepatitis C Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Astellas Pharma US, Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: FA-788-0004
Record Dates: First submitted 2002-10-18; First posted 2002-10-24 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Hepatitis C
Keywords: HCV
MeSH Terms: conditions — Hepatitis C

INTERVENTIONS:
Drug: FK788

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of 4 weeks therapy with FK788 in subjects with chronic hepatitis C virus (HCV) infection. Also, to assess the effect of FK788 on serum ALT concentration and hepatitis C viral level during therapy and for four weeks following therapy.

DETAILED DESCRIPTION:
This is a multi-center, randomized, investigator and subject blinded, placebo-controlled eight week study, including a four week treatment period and a four week follow-up period. Three cohorts of HCV positive subjects will be studied in a sequential manner.

ELIGIBILITY:
The following criteria is a brief summary of Criterion required for trial participation.

Inclusion Criteria

* Has chronic hepatitis C virus infection and has previously received at least three months of treatment with any approved therapy and failed to respond, relapsed or did not tolerate therapy
* Has positive HCV RNA by RT-PCR
* Has abnormal ALT levels (at least 2 X ULN)
* Has liver biopsy within past 2 years consistent with chronic hepatitis, no evidence of non-alcoholic steatohepatitis or cirrhosis, and at least mild inflammation
* Has normal liver function indicated by: PT =< 2 sec. prolonged compared to the ULN, Albumin >= 3.5 g/dL, Total bilirubin =< 1.5 mg/dL
* ANA titer =< 1:160

Exclusion Criteria

* Has positive skin test for tuberculosis
* Has ALT value >= 300 IU/L
* Has abnormal hematological parameters indicated by: ANC < 1500/mm3 and Platelets < 100,000/mm3
* Has creatinine > 1.5 X ULN
* AFP > 50 ng/mL and evidence of hepatocellular carcinoma on ultrasound
* Is a carrier of the hepatitis B surface antigen (HBsAg), positive for HIV-1 and/or HIV-2 antibodies

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48
Dates: Start 2002-10; Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Liver Center Huntington Memorial Hospital, Pasadena, California
  - Rocky Mount Gastroenterology, Lakewood, Colorado
  - University of Florida and Shands Hospital, Gainsville, Florida
  - Liver Center BIDMC - Harvard, Boston, Massachusetts
  - Gastroenterology and Hepatology, Kansas City, Missouri
  - Carolinas Center for Liver Disease, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Thomas Jefferson University, Gastroenterology and Hepatology, Philadelphia, Pennsylvania
  - Northwest Medical Specialties, PLLC Infections Limited, P.S., Tacoma, Washington